CLINICAL TRIAL: NCT01775605
Title: Randomized Study of the Use of Synera for Pain Relief During Local Lidocaine Needle Skin Infiltration for Epidural Placement in Subjects Undergoing Elective Cesarean Section.
Brief Title: Study of Use of Synera for Pain During Local Skin Infiltration With Lidocaine Before Epidural Placement
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 11-376
Record Dates: First submitted 2012-12-10; First posted 2013-01-25 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Pain; Anxiety
Keywords: Subject
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Synera (Active Comparator): Synera Pain Patch
  Interventions: Drug: Synera
- No patch control (No Intervention): No intervention group
- Control (Sham Comparator): Sham
  Interventions: Drug: Synera

INTERVENTIONS:
Drug: Synera — Synera Pain Patch
  Arms: Control; Synera

SUMMARY:
Local infiltration with lidocaine prior to epidural placement for cesarean section, although brief, can be painful. This pain can lead to increased anxiety and distress, adversely affecting patient's overall experience. This study proposes to examine the application of Synera pain patch prior to lidocaine infiltration to reduce this pain and anxiety.

The primary objective of this study is to determine the effect of the Synera on maternal experience during epidural placement. The efficacy of Synera pain patch in reducing subject pain during skin infiltration with lidocaine prior to epidural placement in subjects presenting for scheduled cesarean section will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Undergoing pre-scheduled cesarean section;
* Expected singleton birth;
* BMI <=35kg.m-2;

Exclusion Criteria:

* Undergoing emergency cesarean section;
* Complications during pregnancy;
* History of hypersensitivity to study medication(lidocaine or tetracaine) or para-aminobenzoic acid;
* Allergies to bird proteins, feathers, or egg products; or any other skin allergies; dermatitis an open wound at the patch site or a history of difficult epidural placement;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rating of pain intensity upon lidocaine infiltration | 30 minutes (following patch placement , upon lidocaine infiltration)

SECONDARY OUTCOMES:
Subject anxiety | 1 hour (Upon admission to surgical holding area and after epidural placement)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Strobel, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore Unniversity Hospital, Manhasset, New York, United States